CLINICAL TRIAL: NCT03389633
Title: Does Cardiac Rehabilitation Reduce the Risk of Recurrence of Atrial Fibrillation Following the First Catheter Ablation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: prof. dr. Paul Dendale (Other)
Responsible Party: Sponsor-Investigator, prof. dr. Paul Dendale, Professor of cardiovascular pathophysiology, Hasselt University
Organization: Hasselt University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16.46/cardio16.08
Record Dates: First submitted 2017-12-20; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation group (Experimental): this group follows a 3 months rehab program
  Interventions: Other: rehabilitation
- No rehabilitation (No Intervention): This group does not follow a rehab program

INTERVENTIONS:
Other: rehabilitation
  Arms: Rehabilitation group

SUMMARY:
Many risk factors contribute to the onset of atrial fibrillation. This study is specifically concerned with the effect of addressing these risk factors by cardiac rehabilitation on the risk of recurrence of atrial fibrillation following catheter ablation. A non-randomized, retrospective study was performed on patients treated with a catheter ablation for atrial fibrillation. The intervention group consisted of patients who chose to participate in the cardiac rehabilitation program. The control group only received standard care. The primary objective was to examine whether cardiac rehabilitation following the first ablation for atrial fibrillation resulted in a reduction of the time to or the risk of recurrence of atrial fibrillation or the need for a second ablation within 1 year after the first ablation. A Kaplan-Meier analysis was used to examine the primary objective. The secondary objectives of this study were to examine whether cardiac rehabilitation following the first ablation for atrial fibrillation had an effect on the evolution of the patients' BMI (a Mann-Whitney U test), the number of recurrences of atrial fibrillation (a Poisson regression) and the proportion of patients who need to continue treatment with antiarrhythmics 3 months following the first ablation (a chi-square test).

DETAILED DESCRIPTION:
The intervention group follows a 3 months rehab program consisting of training, education, coaching and medical follow-up. The control group are patients that chose not to follow this program. This is a retrospective non randomized trial

ELIGIBILITY:
Inclusion Criteria:

* an ablation for AF (Atrial fibrillation)

Exclusion Criteria:

* a complicated ablation
* a prosthetic heart valve
* a severe valvulopathy,
* hyperthyroidism at the time of the ablation,
* pregnancy and breastfeeding,
* intensive sport (more than 1 hour a day),
* a myocardial infarction or a thromboembolic event within 3 months after the ablation,
* a pacemaker
* end-stage renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Number of recurrences of atrial fibrillation or need for new ablation | from 3 months after discharge until 1 year
  idem

SECONDARY OUTCOMES:
The proportion of patients who needed to continue treatment with antiarrhythmics | month 3 until one year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dendale, prof. dr., Principal Investigator — Jessa Hospital

IPD SHARING:
Plan to Share IPD: Undecided